CLINICAL TRIAL: NCT00803322
Title: Community Health Workers Improve Tuberculosis Case Notification and Treatment Success in Southern Ethiopia
Brief Title: Improving Community Based Tuberculosis Care in Ethiopia
Acronym: community
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Centre for International Health, SNNP Regional health Bureau (Unknown)
Responsible Party: Daniel Gemechu Datiko, Centre for International Health, SNNP Regional health Bureau
Other Study IDs: 0001; 001
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Pulmonary Tuberculosis
Keywords: TB; community; community health workers; Ethiopia; identify suspects of pulmonary tuberculosis; collect sputum specimen for examination; treat smear positive cases in the community
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: communities where tuberculosis patients followed the conventional health facility based tuberculosis case finding and treatment
- 2: community where suspects of pulmonary tuberculosis were identified by community health workers and received treatment in the community

SUMMARY:
The purpose of this study is to see if involving community health workers improves tuberculosis case finding and treatment outcome.

DETAILED DESCRIPTION:
Tuberculosis suspects in the study area

Outcome smear positive tuberculosis cases identified smear positive tuberculosis cases treated

ELIGIBILITY:
Inclusion Criteria:

* suspects of pulmonary tuberculosis

Exclusion Criteria:

* not in the study area

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: suspects of pulmonary tuberculosis in the study are. In group two suspects were identified and treated bo community health workers while in group on used the conventional health facility based tuberculosis diagnosis and treatment
Sampling Method: Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
smear positive tuberculosis case notification rate | september 2006 - setmeber 2007

SECONDARY OUTCOMES:
smear positive treatment success rate | september 2006 - April 2007

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Datiko, MD, Principal Investigator — CIH of Bergen University and RHB of SNNPRS Ethiopia; Bernt Lindtjorn, Study Director — CIH UIB
Locations (1):
- Dale and Wonsho districts Sidama zone, Southern Ethiopia, Irgalem, Snnpr, Ethiopia

REFERENCES:
- [Derived] Datiko DG, Lindtjorn B. Cost and cost-effectiveness of smear-positive tuberculosis treatment by Health Extension Workers in Southern Ethiopia: a community randomized trial. PLoS One. 2010 Feb 17;5(2):e9158. doi: 10.1371/journal.pone.0009158. PMID 20174642
- [Derived] Datiko DG, Lindtjorn B. Health extension workers improve tuberculosis case detection and treatment success in southern Ethiopia: a community randomized trial. PLoS One. 2009;4(5):e5443. doi: 10.1371/journal.pone.0005443. Epub 2009 May 8. PMID 19424460